CLINICAL TRIAL: NCT07339839
Title: Glecirasib Combined With Ivonescimab for First-line Treatment of KRAS G12C-mutated Locally Advanced or Metastatic Non-Small Cell Lung Cancer: A Prospective, Multi-center, Phase I/II Clinical Study
Brief Title: Glecirasib Combined With Ivonescimab for First-line Treatment of KRAS G12C-mutated NSCLC
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zhijie Wang, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC5886
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: NSCLC Stage IV; KRAS G12C
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glecirasib Combined With Ivonescimab (Experimental)
  Interventions: Drug: Glecirasib; Drug: Ivonescimab

INTERVENTIONS:
Drug: Glecirasib — For Phase I Dose Escalation, Glecirasib includes 2 dose cohorts: 600 mg QD and 800 mg QD, respectively, to determine the Glecirasib PR2D dose for the Phase II study.
  Other Names: JAB-21822
Drug: Ivonescimab — Administered intravenously at 20 mg/kg, every 3 weeks (Q3W).
  Other Names: AK112

SUMMARY:
This study evaluates the safety, tolerability, maximum tolerated dose (MTD), dose-limiting toxicities (DLTs), and recommended phase II dose (RP2D) of Glecirasib in combination with Ivonescimab in patients with previously untreated, KRAS G12C-mutated, locally advanced or metastatic non-small cell lung cancer (NSCLC) with PD-L1 TPS ≥1%. The study includes a Phase I 3+3 dose-escalation stage followed by a Phase II Simon two-stage design to assess preliminary antitumor efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Age ≥18 years.
* Newly diagnosed, unresectable, locally advanced (ineligible for curative concurrent - chemoradiotherapy) or metastatic NSCLC per AJCC 9th edition.
* KRAS G12C mutation confirmed by validated testing.
* PD-L1 TPS ≥1%.
* ≥1 measurable lesion per RECIST v1.1.
* No prior systemic therapy for advanced/metastatic NSCLC; prior adjuvant therapy allowed if completed >6 months before dosing and toxicities recovered to ≤Grade 1.
* ECOG PS 0-2.
* Life expectancy >3 months
* Adequate organ function (hematologic, hepatic, renal, coagulation per protocol thresholds)
* Negative pregnancy test for women of childbearing potential; adequate contraception for men and women through 3 months post-treatment
* Willing and able to comply with study procedures and follow-up.

Exclusion Criteria:

* History of other malignancies (exceptions: cured basal cell carcinoma, cervical carcinoma in situ)
* Predominant squamous NSCLC, small cell carcinoma, or neuroendocrine carcinoma.
* Other actionable drivers (EGFR, ALK, ROS1, RET, BRAF, NTRK, MET, etc.).
* Known hypersensitivity to study drugs.
* Prior PD-1/PD-L1 inhibitors or KRAS inhibitors.
* Active autoimmune disease or autoimmune disease history requiring systemic therapy.
* Systemic immunosuppressive therapy within 14 days prior to first dose.
* Symptomatic ascites/pleural effusion needing recurrent drainage.
* Significant cardiovascular disease (NYHA ≥2, MI within 1 year, uncontrolled arrhythmias).
* Active infection, unexplained fever >38.5°C.
* Interstitial lung disease or pneumonitis.
* HIV infection or other immunodeficiency.
* Live vaccines within 4 weeks.
* Substance abuse, alcoholism, or psychiatric disorders impairing compliance.
* Unable to swallow oral medication.
* Any condition that may interfere with study participation or interpretation as judged by investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Phase I: Maximum Tolerated Dose (MTD) | 21 days after the first dose.
  The MTD is determined using a standard 3+3 dose-escalation design. It is defined as the dose level prior to the dose at which ≥2 out of 3-6 patients experience a Dose-Limiting Toxicity (DLT) within the first 21 days of treatment
Phase I: Incidence of Dose-Limiting Toxicities (DLTs) | 21 days after the first dose.
  Evaluation of toxicities related to the study drugs, including hematologic and non-hematologic toxicities as defined in the protocol.
Phase I: Recommended Phase 2 Dose (RP2D) | 21 days after the first dose.
  The RP2D of Glecirasib in combination with Ivonescimab will be selected based on the comprehensive evaluation of the MTD, DLT occurrences, and overall safety data observed during the Phase I escalation phase. This dose will then be utilized in the Phase II Simon's two-stage expansion to further evaluate efficacy and safety.
Phase II: Objective Response Rate (ORR) | Assessed up to 24 months
  The proportion of patients who achieve a Complete Response (CR) or Partial Response (PR) based on RECIST v1.1.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Up to 24 months
  Proportion of patients with CR, PR, or SD.
Progression-Free Survival (PFS) | Up to 24 months
  Time from the first dose to the first documented disease progression or death from any cause.
Duration of Response (DOR) | Up to 24 months
  Time from the first documented response (CR or PR) to progression or death.
Overall Survival (OS) | Up to 24 months
  Time from the first dose to death from any cause
Incidence of Adverse Events (AEs) | From first dose enrollment through 28 days after the last dose.
  Severity of AEs graded by CTCAE v5.0

IPD SHARING:
Plan to Share IPD: No